CLINICAL TRIAL: NCT05004298
Title: Evaluation of an Animal Assisted Therapy Program in People With Mental Illness, for the Promotion of Positive Mental Health Behaviors
Brief Title: Evaluation of an Animal Assisted Therapy Program in People With Mental Illness, and Promotion of Positive Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIBSP-TAA-2020-122
Record Dates: First submitted 2021-07-18; First posted 2021-08-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-09

CONDITIONS: Mental Disorders, Severe
Keywords: Positive Mental Health; Mental Illness,; Animal Assisted Therapy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animal assisted terapy (Experimental): The Experimental Group, in addition to receiving the usual activities of the rehabilitation device. You will receive the ten weekly sessions of the TAA Program.The program structure will aim to influence the 6 specific factors, described in the Multifactorial Model of Positive Mental Health of Dr. Lluch, which are: F1-Personal Satisfaction, F2-Prosocial Attitude, F3-Self-control, F4-Autonomy, F5- Problem Solving and Self-actualization and F6 Interpersonal Relationship Skills. For this reason, direct contact exercises with the dog will be designed and defined to work on them.
  Interventions: Other: Animal Assited therapy
- Control Group (No Intervention): The Control Group will receive the usual activities of the rehabilitation device.

INTERVENTIONS:
Other: Animal Assited therapy — The intervention will be structured in 10 group sessions, with a weekly frequency and one hour duration.
  Arms: Animal assisted terapy

SUMMARY:
Scientific literature reports that focusing interventions on people with mental health problems, from the threshold of Positive Mental Health, is effective and allows the person to promote positive mental health behaviors. The well-known Animal Assisted Therapy is a complementary intervention used for decades that has reported scientific evidence in the field of mental health in communication, socialization, anxiety and adherence to treatment of patients.

This protocol aims to create and evaluate an Assisted Therapy program with dogs in relation to the development and promotion of Positive Mental Health behaviors in people with mental illness in a community rehabilitation service.

DETAILED DESCRIPTION:
Background Mental health problems have a high prevalence. According to data provided by the World Health Organization (WHO), one in four people will suffer from some form of lifelong mental health problem and it is estimated that some 450 million people currently suffer from it. These are disorders that generate a social, economic and family burden that is expected to increase significantly over the next 20 years.

"Contribute to the promotion of positive mental health and well-being of people throughout their lives by developing specific programs for people with mental disorders, adapted to each stage of life and based on the promotion of healthy habits in physical, cognitive and emotional health ", is the first strategic line proposed by the European Mental Health Action Plan 2013/2020 (EMHAP).

In Catalonia, with the same approach, the strategies of the "Master Plan for Mental Health and Addictions 2017/2020" are elaborated whose objective is the promotion of health and prevention of the disease, all this, with a community base that prioritizes the recovery of the person oriented towards social and labor inclusion, and improve their quality of life.

The field of mental health intervention has changed its paradigm and approach. Since the middle of the twentieth century, a change has been looming, not only in the treatment of the disorder itself, but also in its prevention. Despite this change, the reality is that it is still, in many cases in mental health centers, mainly involved in the field of mental illness and clinical symptoms. It is relevant that interventions for people with mental health problems are attractive, to encourage commitment and with a positive approach, from the threshold of Positive Mental Health (PMH)) .

The term PMH itself, focuses on understanding the mental functioning of human beings from a "positive" perspective, ie, healthy, optimistic, oriented to well-being and personal growth.

Lluch, mention in their chapter, that interventions must be performed from a positive perspective, based on healthy actions with actions that help strengthen and enhance the level of mental health.

The literature describes two models for framing the concept of PMH on the one hand, in 1958, the Jahoda PMH model and on the other hand in 1999, the Lluch´s Multifactorial PMH Model.

To implement this new vision of the care model, aimed at promoting and preventing mental health in people with these disorders, new alternative and non-pharmacological strategies and programs are framed to develop PMH behaviors. One of these interventions is known as Animal Assisted Therapy (AAT).

The scientific literature reports multiple benefits of AAT in the field of mental health, one of which focuses on the influence on socialization as an effect of interaction with the animal. At York Hospital, England, therapeutic contact with small farm animals was introduced in order to promote self-control. In the twentieth century in the United States, this animal therapy was applied in the treatment of hospitalized adults and children in order to improve their quality of life .

Morris reviewed published scientific studies between 1996 and 2006 on the effects of AATs. In this review he proposed the use of AATs at any age, in any field of action and with people in need of improving their mood, motivation, self-esteem and sense of well-being.

Bert, conducted a systematic review of the benefits of AATs. Of the 36 selected studies, five were performed in the field of psychiatry. Most studies included dogs. The authors concluded that AATs provide benefits, such as reducing stress, pain, and anxiety. Changes in vital signs and nutritional intake were also reported as a result.

Calvo, in their 24-week study of AAT with adults and mental illness, reported benefits in relation to negative symptoms, increased adherence to the therapeutic program, and reduction of post-session cortisol.

There are several authors who highlight the definition of assisted therapy with animals, Vallejo in 2006, defines AAT as those methods that include human interaction with animals in prevention and treatment of human pathologies, both physical and mental, that is, animal-assisted therapy is performed when a human interacts with the animal under predetermined therapeutic criteria in those therapies that are intended to solve certain health disorders. This intervention has predesigned goals in order to obtain physical, social, emotional and cognitive therapy benefits in a variety of pathologies, such as schizophrenia, conduct disorders, Down Syndrome and autism, among others .

Jones, in relation to the incorporation of animal-assisted therapy in mental health treatments for adolescents, 7 studies were examined, the common objective of all of them was to reduce the impact of psychological disorders to improve functioning and functioning. adolescent adaptation.

Stefanini, in 2015, randomly applied AAT to 34 hospitalized adolescent patients, who presented acute psychiatric pathology, and their evolution was compared with a control group. The treatment consisted of weekly therapy sessions lasting 45 minutes, for three months. The results highlighted an improvement in clinical evolution and recovery, as well as an improvement in emotional and behavioral symptoms and in their global competence.

This protocol aims to create and evaluate an Assisted Therapy program with dogs in relation to the development and promotion of Positive Mental Health behaviors in people with mental illness in a community rehabilitation service.

Hypothesis People diagnosed with a mental disorder who participate in the AAT program with dogs will exhibit behaviors, with a higher level of PMH, than before the intervention.

Method / Design Mixed study with two phases. A first qualitative phase, with a focus group, which will analyze the validity of the intervention. In the second phase, a pre-experimental design is proposed, post-test test of a single group, after the intervention of Animal Assisted Therapy.

General objective, phase I. To analyze the validity of a Assisted Therapy program with dogs, aimed at people with mental illnesss.

General objective, phase II. The overall goal is to evaluate the effectiveness of AAT intervention with dogs.

Data collection will be done through an ad hoc form and the Lluch Positive Mental Health Questionnaire (1999).

Definition of variables For phase I, structural variables are defined around which the interview guide will be elaborated: 1) Relevance of the interventions / activities proposed in the program, 2) Conceptual composition of the sessions with practical application of the 6 specific factors of PMH of the Lluch Multifactorial Model, 3) Criteria for selecting participants, 4) Procedure for implementing the program, 5) Duration of the sessions.

For the second phase, that of the intervention, in itself, are defined:

Socio-demographic variables: 1) Age, 2) Sex, 3) Nationality, 4) City of residence, 5) Level of education, 6) Number of siblings, 7) Guardianship by Foundation, 8) Maintaining contact with family, 9) People with which he usually lives, 10) Having previously had contact with animals at the family level (Only for phase II-B).

Health variables: 1) Affiliated psychiatric diagnosis, 2) Medical treatment performed, 3) Pharmacological treatment performed, 4) Tobacco use, 5) Number of cigarettes per day, 6) Alcohol consumption, 7) Consumption of other toxic substances.

Socio-demographic and health variables will be measured before the start of the first session of the intervention.

Independent variable: The animal-assisted intervention program itself, intervention program will be structured in 10 sessions with a weekly frequency and a duration of 1 hour Dependent variables: The variables in this section were defined through Lluch's (1999) Multifactorial Positive Mental Health Model which consists of 6 PMH-specific factors, and together with the global analysis of the construct, form a total of 7 variables: 1) Global PMH Level, 2) PMH Level in each of the 6 Model Specific Factors: F1) Personal Satisfaction, F2) Prosocial Attitude, F3) Self-Control, F4) Autonomy, F5) Problem Solving and Self-Update, F6 ) Interpersonal Relationship Skills6. The variable will be measured before the start of the first session of the intervention and after the last session of the same.

Expected sample size For this study, three groups of experts consisting of 8 people will be created. For the intervention phase. The department has 100 places for people with mental illness. Professionals, through non-probabilistic convenience sampling, will include participants as users attend a follow-up visit with a nurse, meet established criteria, and accept their participation. It is contemplated to include in this phase those people linked during the 12 months from the beginning of the intervention. It is planned to recruit 30 cases in the planned period.

Data Management and Analysis For the second phase, an initial descriptive analysis of the sociodemographic, health and quantitative variables will be performed. For this, measures of central tendency and dispersion will be used, for the quantitative variables (mean and standard deviation). For the analysis of the categorical variables, the number of cases (absolute frequency) as well as the percentage will be provided. 95% confidence intervals will be calculated for both measurements and percentages (relative frequency).

95% confidence intervals will be calculated for the main variables of interest. For the bivariate analysis the Pearson Square Chi test will be used for the categorical variables. For these in the analysis of paired data, the McNemar test will be taken as a reference.

For the analysis of the association between the quantitative and categorical variables of two levels of repeated measurements, it will be analyzed by the non-parametric Wilcoxon Ranges test, or the "t" test of paired data, in case of related data.

The statistical program chosen for the data analysis will be the Statistical Package for Social Sciences Version 26.0 package.

The results of this study will provide evidence of the effectiveness of an animal-assisted intervention designed from a new intervention paradigm from a positive approach, using the theoretical model of Positive Mental Health. If its effectiveness is proven and the results are acceptable, this could be an innovative strategy for interventions offered in the field of mental health, as it strengthens people's strengths.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with a mental disorder
* Presence of social dysfunction
* Over 18 years
* Voluntary acceptance to the study

Exclusion Criteria:

* Allergies to dogs
* Phobia of dogs
* History of animal abuse
* People whose cognitive capacity does not allow them to follow the sessions of the intervention program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Positive Mental Health Questionnaire Lluch (39-156points) | Data collection will be done using an ad hoc form and the Positive Mental Health Questionnaire Lluch (1999). There is an interval of ten weeks between the pretest and posttest collection.
  Evaluate the effectiveness of the Animal Assisted Therapy Program

CONTACTS AND LOCATIONS:
Overall Officials: Judith Balaguer, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital De la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] World Health Organization (WHO). World Health Organization, Calouste Gulbenkian Foundation. Social determinants of mental health. Geneva [Internet]. 2014; Available from: http://apps.who.int/iris/bitstream/10665/112828/1/9789241506809_eng.pdf?ua=1
- [Result] World Health Organization (WHO). The European mental health action plan 2013-2020. Copenhagen [Internet]. 2015; Available from: http://www.euro.who.int/__data/assets/pdf_file/0020/280604/WHO-Europe-Mental-HealthAcion-Plan-2013-2020.pdf
- [Result] Generalitat de Catalunya. Pla director de salut mental i addiccions 2017-2020.Barcelona: Departament de Salut. 2017; Available from: https://salutweb.gencat.cat/web/.content/_ambits-actuacio/Linies-dactuacio/Estrategies-de-salut/Salut-mental-addiccions/Linies-estrategiques/estrategies2017_2020.pdf
- [Result] Lluch MT. Concepto de salud mental positiva: factores relacionados. En: Fornés-Vives J, Gómez-Salgado J, eds. Recursos y programas para la salud mental : enfermería psicosocial II. Madrid: Funden. 2008;37-69.
- [Result] Mission Australia in association with Black Dog Institute. Youth Mental Health Report: Youth Survey 2012-16. 2016;5-21. Available from: https://www.missionaustralia.com.au/publications/...mental-health-youth-report/file
- [Result] Fernandez Alonso MC, Buitrago Ramirez F, Ciurana Misol R, Chocron Bentata L, Garcia Campayo J, Monton Franco C, Tizon Garcia JL; Grupo de Salud Mental del PAPPS. [Prevention of mental health disorders]. Aten Primaria. 2012 Jun;44 Suppl 1(Suppl 1):52-6. doi: 10.1016/S0212-6567(12)70014-8. No abstract available. Spanish. PMID 23399507
- [Result] Lluch MT, Sequeira C, J R. La salud mental positiva desde una perspectiva multifactorial. In En V. Fragoso y M. Sotto Mayor (Coords.), Gerontologia e transdisciplinariedade I (pp. 114-129). Sâo Paulo (Brasil): Portal Ediçôes Envelhecimento; 2017.
- [Result] Jahoda M. Current concepts of positive mental health. New York: Basic Books. 1958;
- [Result] Lluch T. Evaluación empírica de un modelo conceptual de salud mental positiva. Salud Ment. 2002;25(4):42-55.
- [Result] Lluch MT. Construcción y análisis psicométrico de un cuestionario para evaluar la salud mental positiva. Rev Int Psicol clínica y la salud. 2003;1:61-78.
- [Result] Sánchez-Ortega MA, Puig-Llobet M, Lluch-Canut MT. Efectividad de un programa de intervención psicosocial enfermera para potenciar la agencia de autocuidado y la salud mental positiva en personas con problemas crónicos de salud. 2010;326. Available from: http://diposit.ub.edu/dspace/bitstream/2445/101363/1/MASO_TESIS.pdf
- [Result] Sanromà Ortiz M. Evaluación de un programa de empoderamiento para potenciar y desarrollar conductas promotoras de salud y salud mental positiva en estudiantes de enfermería. "Dinamiza la Salud: Cuídate y Cuida ". TDX (Tesis Dr en Xarxa) [Internet]. 2016 Apr 26 [cited 2020 May 18]; Available from: http://www.tdx.cat/handle/10803/386481
- [Result] Amar J, Palacio J, Norte U, Llinás H, Puerta L, Sierra E, et al. Calidad de vida y Salud Mental Positiva en Menores Trabajadores De Toluviejo. Suma Psicológica. 2008;15(2):385-403.
- [Result] Fine AH. Handbook on Animal-Assisted Therapy: Theoretical Foundations and Guidelines for Practice. 3rd ed. Academic Press; 2010. 588 p.
- [Result] Calvo P, Fortuny JR, Guzman S, Macias C, Bowen J, Garcia ML, Orejas O, Molins F, Tvarijonaviciute A, Ceron JJ, Bulbena A, Fatjo J. Animal Assisted Therapy (AAT) Program As a Useful Adjunct to Conventional Psychosocial Rehabilitation for Patients with Schizophrenia: Results of a Small-scale Randomized Controlled Trial. Front Psychol. 2016 May 6;7:631. doi: 10.3389/fpsyg.2016.00631. eCollection 2016. PMID 27199859
- [Result] Olarte MA, Díaz VM. Intervenciones asistidas por animales: Intervenciones con perros en adultos mayores a partir del enfoque multimodal. Rev científica Eur [Internet]. 2016;5(10):269-86. Available from: https://doi.org/10.19044/esj.2016.v12n10p%25p
- [Result] Martínez R. La terapia asistida por animales: Una perspectiva y línea de investigación en la atención a la diversidad. Indivisa Bol Estud Investig. 2008;9:117-44
- [Result] Morris SB. Estimating effect sizes from pretest-posttest-control group designs. Org Res Methods. 2007;11:364-386
- [Result] Bert F, Gualano MR, Camussi E, Pieve G, Voglino G, Siliquini R. Animal assisted intervention: A systematic review of benefits and risks. Eur J Integr Med. 2016 Oct;8(5):695-706. doi: 10.1016/j.eujim.2016.05.005. Epub 2016 May 20. PMID 32362955
- [Result] Cabra C. Terapia asistida con animales. Efectos positivos en la salud humana. J Agric Anim Sci. 2012;1(2):32-45.
- [Result] Vallejo R. Introducción a la psicopatología y a la Psiquiátria. Sexta edic. Barcelona, España: Elsevier; 2006. 344 p
- [Result] Alonso Y. ¿Los animales fomentan la salud humana? Un análisis preliminar. Rev.de Psicol Gral y Aplic. 2000;53(4):693-700.
- [Result] Oropesa, P., Wilson, I.G., Saní, M., Gaínza Y. Terapia asistida con animales como fuente de recurso en el tratamiento rehabilitador. Medisan [Internet]. 2009;0-0. Available from: http://www.redalyc.org/articulo.oa?id=368448456014%0A
- [Result] Jones MG, Rice SM, Cotton SM. Incorporating animal-assisted therapy in mental health treatments for adolescents: A systematic review of canine assisted psychotherapy. PLoS One. 2019 Jan 17;14(1):e0210761. doi: 10.1371/journal.pone.0210761. eCollection 2019. PMID 30653587
- [Result] Stefanini MC, Martino A, Allori P, Galeotti F, Tani F. The use of Animal-Assisted Therapy in adolescents with acute mental disorders: A randomized controlled study. Complement Ther Clin Pract. 2015 Feb;21(1):42-6. doi: 10.1016/j.ctcp.2015.01.001. Epub 2015 Jan 29. PMID 25701449
- [Result] Stefanini MC, Martino A, Bacci B, Tani F. The effect of animal-assisted therapy on emotional and behavioral symptoms in children and adolescents hospitalized for acute mental disorders. Eur J Integr Med [Internet]. 2016;8(2):81-8. Available from: http://dx.doi.org/10.1016/j.eujim.2016.03.001